CLINICAL TRIAL: NCT00283413
Title: Symbiot III: A Prospective Randomized Trial Evaluating the Symbiot Covered Stent System in Saphenous Vein Grafts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Matthew Albert/Clinical Project Manager, Boston Scientific Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G980213; S2001
Record Dates: First submitted 2006-01-27; First posted 2006-01-30 (Estimated); Last update posted 2009-11-02 (Estimated); Status verified 2009-10

CONDITIONS: Symptomatic Ischemic Saphenous Vein Graft Disease
Keywords: Covered Stent System; Saphenous Vein Graft; Coronary Artery Bypass[MeSH]; Stents[MeSH]

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Symbiot Covered Stent System
  Interventions: Device: Covered Stent System
- 2 (Active Comparator): Commercially available bare metal stent
  Interventions: Device: Bare metal stent

INTERVENTIONS:
Device: Covered Stent System — Self-expanding, polytetrafluoroethylene(PTFE)-covered, stent system
  Other Names: Symbiot Covered Stent System
  Arms: 1
Device: Bare metal stent — Any commercially available bare metal stent for coronary indication
  Arms: 2

SUMMARY:
The objective of the Symbiot III Clinical Trial was to evaluate the safety and effectiveness of the Symbiot Covered Stent System in the treatment of symptomatic ischemic saphenous vein bypass graft disease.

DETAILED DESCRIPTION:
Symbiot III was a prospective, multi-center, randomized, controlled trial to evaluate the safety and efficacy of the Symbiot stent compared to bare metal stents in the treatment of symptomatic ischemic saphenous vein graft disease. Randomization was stratified by the intended use of intravenous glycoprotein IIb/IIIa inhibitors and by the intended use of approved distal protection to ensure approximate balance between study treatments within each of the strata. The primary outcome variable for the study was target lesion percent diameter stenosis at 8 months post-implant.

ELIGIBILITY:
General Inclusion Criteria:

1. Patient >=18 years old
2. Patients is eligible for percutaneous coronary intervention and stenting
3. Patient is an acceptable candidate for repeat CABG
4. CPK must be within ULN on the day of the procedure
5. Patient must meet one of the following requirements:

   * treatment of one or two de novo or restenotic lesions in a single SVG
   * treatment of both a native coronary artery and the target graft in a single procedure, provided that the native artery is treated prior to randomization of the target lesion(s) and did not result in MACE or TIMI flow <3
6. Patients (or their legal representative) understands the nature of the procedure and study requirements and provides written informed consent before any study specific tests or procedures are performed
7. Patient is willing to comply with specified follow-up evaluations at the specified times and locations
8. Patient has angina pectoris (CCS 1, 2, 3, or 4) or coronary ischemia documented by a positive functional ischemia study
9. Patient has no child bearing potential or has a negative pregnancy test within 7 days prior to treatment

Angiographic Inclusion Criteria:

1. Target lesion(s) are located within a single SVG
2. Reference vessel >=3.5 mm and <=5.5mm in diameter at the stent deployment site
3. Cumulative target lesion length is <=41mm
4. Target lesion(s) randomized to treatment with the study device must be completely covered by 1 or 2 stents (maximum allowable aggregate stent length in target vessel of 51 mm)
5. Target lesion stenosis >=50% and <100%

General Exclusion Criteria:

1. Patient is currently enrolled in another IRB-approved trial that has not reached the primary endpoint visit or is still in the active treatment phase
2. Patient has been previously enrolled in any Symbiot Trial
3. Patient has documented left ventricular ejection fraction of <30% within 30 days of enrollment
4. Patient has had a myocardial infarction within 48 hours prior to trial procedure and/or CK-MB >2X the ULN
5. Patient has had, or will have, a planned additional interventional procedure to any coronary vessel (coronary artery or saphenous vein graft) that does not meet the following criteria:

   If the staged procedure is chosen for non-study percutaneous intervention to any non-target vessel:
   * 30 days or more prior to the index procedure is allowed
   * Between 24 hours and 30 days prior to the index procedure is allowed provided that no major adverse cardiac events resulted from the staged non-study procedure
   * Within 24 hours prior to the index procedure not allowed
   * Within 30 days after the index procedure is not allowed
   * 30 days or more after the index procedure is allowed
6. The lesion to be treated is within 10 mm of any anastomosis
7. Patient has life expectancy of less than 1 year due to other medical conditions
8. The lesion(s) to be treated requires debulking prior to stent placement
9. Patient has a pre-existing condition for which aspirin is contraindicated
10. Patient has a pre-existing condition for which clopidogrel and ticlopidine are contraindicated
11. Patient has a known hypersensitivity to nickel

Angiographic Exclusion Criteria:

1. Target vessel is a left main artery-equivalent graft
2. Target vessel is an internal mammary artery graft
3. Target lesion(s) have any intraluminal thrombus present with TIMI flow <3
4. Target vessel has excessive tortuousity unsuitable for delivery and deployment of Symbiot
5. Target lesion(s) is/are within a previous stented segment
6. Target or non-target vessel requires pre-treatment with an adjunctive non-balloon device (e.g., DCA, TEC, Rotablator or laser) prior to stent placement during the stent placement procedure
7. Treatment with non-approved distal protection systems
8. Target lesion(s) involve either the ostium or distal anastomosis
9. Target lesion(s) are at or immediately distal to a >45 degree bend in the vessel
10. Target vessel is a degenerated SVG (diffuse segments of disease >41 mm in length with stenosis, ectasia and probable thrombus)
11. Untreated lesions are present proximal or distal to the target site which may compromise inflow or outflow of the treatment site after stent deployment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2002-03; Primary Completion 2004-05 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Percent diameter stenosis at 8 months post-implant | 8 Months

SECONDARY OUTCOMES:
Major adverse cardiac event rate at 30 days post-implant | 30 Days

CONTACTS AND LOCATIONS:
Overall Officials: Mark Turco, MD, Principal Investigator — Washington Adventist Hospital, Takoma Park, MD; Maurice Buchbinder, MD, Principal Investigator — Foundation for Cardiovascular Medicine, La Jolla, CA
Locations (49):
- United States (47):
  - Baptist Medical Center Princeton, Birmingham, Alabama
  - University of Alabama Hospital, Birmingham, Alabama
  - Baptist Medical Center South, Montgomery, Alabama
  - Arizona Heart Institute, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - St. Agnes Medical Center, Fresno, California
  - Glendale Memorial Hospital, Glendale, California
  - Scripps Memorial Hospital, La Jolla, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mercy General Hospital, Sacramento, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Palm Beach Heart Research Institute, Atlantis, Florida
  - Munroe Regional Medical Center, Ocala, Florida
  - Florida Hospital, Orlando, Florida
  - University Community Hospital, Tampa, Florida
  - Medical Center of Central Georgia, Macon, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - Methodist Hospital, Indianapolis, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Jewish Hospital & St. Mary's Healthcare, Louisville, Kentucky
  - Maine Medical Center, Portland, Maine
  - Washington Adventist Hospital, Takoma Park, Maryland
  - St. Joseph Medical Center, Towson, Maryland
  - St. John Hospital & Medical Center, Detroit, Michigan
  - Cardiac & Vascular Research Center of Northern Michigan, Petoskey, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - St. Luke's Hospital, Kansas City, Missouri
  - Lenox Hill Hospital, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - Presbyterian Healthcare, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Medical Center, Raleigh, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Providence Hospital, Columbia, South Carolina
  - Memorial Hospital, Chattanooga, Tennessee
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Covenant Medical Center, Lubbock, Texas
  - Baptist Medical Center, San Antonio, Texas
  - Fletcher Allen Health Care, Burlington, Vermont
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Sacred Heart Medical Center, Spokane, Washington
  - Charleston Area Medical Center, Charleston, West Virginia
  - St. Luke's Medical Center, Milwaukee, Wisconsin
- Canada (2):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Montreal Heart Institute, Montreal, Quebec

REFERENCES:
- [Result] Turco MA, Buchbinder M, Popma JJ, Weissman NJ, Mann T, Doucet S, Johnson WL Jr, Greenberg JD, Leadley K, Russell ME. Pivotal, randomized U.S. study of the Symbiottrade mark covered stent system in patients with saphenous vein graft disease: eight-month angiographic and clinical results from the Symbiot III trial. Catheter Cardiovasc Interv. 2006 Sep;68(3):379-88. doi: 10.1002/ccd.20873. PMID 16892434